CLINICAL TRIAL: NCT04370366
Title: Imaging Endolymphatic Hydrops at 7T MRI: Validation of Internal Inner Ear Structures on T2w Imaging as Markers of Endolymphatic Hydrops and a Comparison of Diagnostic Outcomes With 3T MRI
Brief Title: Imaging of Endolymphatic Hydrops at 7T MRI
Status: Recruiting | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other); Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 259867
Record Dates: First submitted 2020-04-29; First posted 2020-04-30 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Meniere Disease
MeSH Terms: conditions — Meniere Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Imaging endolymphatic hydrops with 7T Sodium Imaging and 1.5 T gadolinium enhanced imaging: a comparison of diagnostic outcomes with 3T MRI

Duration of study 24 months

Study design Prospective cohort study

Number of patients 16 patients

1. To evaluate whether imaging both 1.5T and 3T have an equivalent performance in terms of diagnosing MD ears with delayed post gadolinium enhanced MRI (applying quantitative and semi-quantitative analysis)
2. To compare the diagnostic performance of Sodium Imaging at 7T (applying semi-quantitative analysis) with that of delayed post gadolinium enhanced 3T MRI in distinguishing symptomatic from asymptomatic Meniere's Disease (MD) ears.

DETAILED DESCRIPTION:
Meniere's Disease is an inner ear disease characterised by progressive, fluctuating hearing loss and dizziness. Pathologically, it is characterised by endolymphatic hydrops. The diagnosis of Meniere's Disease can be elusive since it relies on the subjective reporting of symptoms and there is no definitive diagnostic test. Non-specific symptoms can occur in the early stages of Meniere's Disease and the disease progression can also fluctuate unpredictably. The cochlear and vestibular compartments may be differentially involved so there maybe clinical variability characterised by solely audiological or vestibular symptoms (1).

The structural correlate of MD is endolymphatic hydrops (EH) , in which the central smaller endolymphatic compartment of the inner ear (including the cochlear duct, saccule and utricle) expands into the surrounding peri-lymphatic chambers. Pathological studies of temporal bones in subjects with MD have demonstrated EH in most cases of Meniere's Disease (2) and its presence is required for, the diagnosis of 'certain Meniere's Disease' according to 1995 American Academy of Otolaryngology-Head and Neck Surgery (AAO-HNS) guidelines (3). An accepted in vivo biological marker for endolymphatic hydrops has yet to be established. Recent developments in MRI technology and techniques have however allowed the demonstration of EH and the clinical application of these imaging studies is now being explored.

High resolution T2-weighted sequences are widely used for the demonstration of labyrinthine anatomy and pathology however they are unable to distinguish the endolymphatic from perilymphatic compartments and hence are generally unable to depict endolymphatic hydrops. The potential role of gadolinium in discriminating the endolymphatic chamber alone first became apparent in animal studies, since gadolinium was seen to accumulate in the perilymph but was excluded from the endolymph by the impermeable tight junctions. Intra-tympanic administration of gadolinium was initially explored, whereby high concentrations could enter the labyrinth through round window diffusion, however the evolution of clinically applicable high resolution sequences at 3T has allowed for gadolinium to be administered by the less invasive intravenous route. Delayed (4 hours post administration) gadolinium enhanced high resolution imaging is now used at a number of centres worldwide for the evaluation of Meniere's Disease patients, although acquisition and analysis methods continue to evolve. This is most frequently performed with 3D Fluid Attenuated Inversion Recovery with variable flip angles turbo spin echo sequence (3D SPACE FLAIR) or 3D real inversion recovery sequence (3D real IR. In order to corroborate the diagnosis of MD, the degree of EH in each cochlea and vestibule is semi-quantitatively graded (4,5) using various scales or may be quantitatively analysed by contouring the size of the two compartments. An ipsilateral increase in the perilymphatic enhancement is an additional MRI feature which is used to help distinguish MD ears.

The identification of cochlear or vestibular hydrops by MRI in vivo may support the diagnosis of Meniere's disease in cases with incomplete phenotypes and where there are other diagnostic considerations such as vestibular migraine or autoimmune ear disease. It may also facilitate early identification, thus guiding future treatment options for patients who have traditionally been required to take a watchful waiting approach to see how their symptoms may evolve or "trial-and-error" approach to management. The identification of bilateral endolymphatic hydrops in a patient with unilateral fluctuating aural symptoms might predict future bilateral disease and potentially influence therapeutic approaches. Establishing imaging as a biomarker in Meniere's disease may allow a contribution to diagnostic criteria and to define homogenous cohorts for longitudinal studies of natural history and treatment response.

However there are deficiencies with this MRI approach which we would like to address with an exploratory study of Meniere's disease patients on 1.5T and 7 Tesla MRI:

1. Due to the small size of the inner ear structures being imaged, and the low concentration of gadolinium in the perilymph, 3T MRI is widely considered as being optimal for the diagnosis of MD. This maximises SNR and improves spatial resolution such that small inner ear structures (e.g. the cochlear duct) maybe delineated, improving precision and inter-observer agreement and diagnostic confidence of EH diagnosis. However there are many institutions which only have access to a 1.5-T system and this potentially limits their investigation of pateints with MD, unless patients are referred to another center. A global market analysis of the distribution of MRI scanners demonstrated that in 2019 there was a 71.3% share of 1.5-T scanners (6). Whilst there are some studies demonstrating feasibility of MD diagnosis on 1.5 T systems (7-9) there has been no study directly comparing the two approaches. It is therefore important to perform a study demonstrating equivalence of diagnostic outcomes at 1.5T and 3T.
2. Gadolinium has an excellent safety record when used at low doses (0.1-0.3 mmol/kg) in patients with normal renal function. However, a causative relationship between gadolinium-based contrast agents and nephrogenic systemic fibrosis is described in patients with renal insufficiency, and there is also increasing evidence that they deposit in the human brain after multiple administrations, although the clinical significance of this remains uncertain (10). Therefore the development of non-contrast enhanced MRI technique is of considerable interest.

Whilst previous MRI approaches have concentrated on the difference in permeability to gadolinium to differentiate the endolymphatic and perilymphatic spaces of the inner ear, the difference in sodium concentrations between the two compartments is another differential feature which has not been explored. The perilymph and endolymph have unique ionic compositions suited to their functions in regulating electrochemical impulses necessary for hearing. The endolymph has a concentration of 1mM/l where the perilymph has a concentration of 140 mmol/l. Sodium imaging with MRI can provide quantitative measures of the sodium concentration in tissue (11,12). It utilizes the signal from the sodium nucleus to acquire images of the sodium biodistribution. Due to the low natural abundance of biological sodium, in comparison to water, as well as a rapid quadrupolar relaxation and lower gyromagnetic ratio the signal available is much lower than that of conventional proton MRI. Together, these properties make sodium very difficult to image with adequate signal-to-noise ratio (SNR) and hence it is most applicable to ultra-high-field MRI (7T) given the significant gain in signal strength.

An initial phase of 7T sodium imaging sequence development has been completed but there remain significant challenges to its application in the inner ear and it remains uncertain whether there will be sufficient spatial resolution and SNR, even at 7T. Therefore, the initially application of Sodium Imaging in MD should be in cases where there is known to be a maximal asymmetry in the size of the endolymphatic compartments on previous imaging studies in order to determine feasibility before determining whether it should be applied to a larger cohort. If Sodium Imaging of the inner ears is considered feasible then correlation of the semiquantitative analysis with the clinical diagnosis and with the size of the endolymphatic structures on reference standard delayed post gadolinium inversion recovery 3T MRI sequences would add validation to this approach.

1. To evaluate whether imaging both 1.5T and 3T have an equivalent performance in terms of diagnosing MD ears with delayed post gadolinium enhanced MRI (applying quantitative and semi-quantitative analysis)
2. To compare the diagnostic performance of Sodium Imaging at 7T (applying semi-quantitative analysis) with that of delayed post gadolinium enhanced 3T MRI in distinguishing symptomatic from asymptomatic Meniere's Disease (MD) ears.

ELIGIBILITY:
Inclusion Criteria

* Male or female, 18 years of age or older
* The capacity to understand the patient information sheet and the ability to provide written informed consent
* Unilateral audio-vestibular symptoms which satisfy 2015 Barany criteria for unilateral Meniere's Disease of less than 5 years duration
* Would be offered clinical MRI scanning for confirmation of a Meniere's disease diagnosis as part of standard of care

Exclusion Criteria:

* Standard contraindications to 7T MRI
* Known allergy to Gadolinium contrast
* Calculated GFR < 30 mls/min
* Previous temporal bone surgery or trauma
* Other known temporal bone pathology
* Requirement for early post gadolinium sequences (e.g. autoimmune inner disease as a differential diagnosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Secondary care. Otology and audio-vestibular clinics Guy's and St Thomas' hospital
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
The qualitative asymmetry of perilymphatic enhancement and the quantitative signal intensity ratio of the cochlea with delayed post gadolinium 3T and 1.5T. | 2.5 years
The semi-quantitative scoring of endolymphatic hydrops and the quantitative volume of endolymphatic and perilymphatic structures with delayed post gadolinium 3T and 1.5T. | 2.5 years
Semi-quantitative analysis (including ratios to internal references and the contralateral ear) of the vestibule on Sodium Imaging at 7T | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen EJ Connor, MRCP FRCR, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pyykko I, Nakashima T, Yoshida T, Zou J, Naganawa S. Meniere's disease: a reappraisal supported by a variable latency of symptoms and the MRI visualisation of endolymphatic hydrops. BMJ Open. 2013 Feb 14;3(2):e001555. doi: 10.1136/bmjopen-2012-001555. Print 2013. PMID 23418296
- [Background] Naganawa S, Sugiura M, Kawamura M, Fukatsu H, Sone M, Nakashima T. Imaging of endolymphatic and perilymphatic fluid at 3T after intratympanic administration of gadolinium-diethylene-triamine pentaacetic acid. AJNR Am J Neuroradiol. 2008 Apr;29(4):724-6. doi: 10.3174/ajnr.A0894. Epub 2008 Jan 9. PMID 18184846
- [Background] Barath K, Schuknecht B, Naldi AM, Schrepfer T, Bockisch CJ, Hegemann SC. Detection and grading of endolymphatic hydrops in Meniere disease using MR imaging. AJNR Am J Neuroradiol. 2014 Jul;35(7):1387-92. doi: 10.3174/ajnr.A3856. Epub 2014 Feb 13. PMID 24524921
- [Background] Attye A, Eliezer M, Boudiaf N, Tropres I, Chechin D, Schmerber S, Dumas G, Krainik A. MRI of endolymphatic hydrops in patients with Meniere's disease: a case-controlled study with a simplified classification based on saccular morphology. Eur Radiol. 2017 Aug;27(8):3138-3146. doi: 10.1007/s00330-016-4701-z. Epub 2016 Dec 20. PMID 27999985
- [Background] Venkatasamy A, Veillon F, Fleury A, Eliezer M, Abu Eid M, Romain B, Vuong H, Rohmer D, Charpiot A, Sick H, Riehm S. Imaging of the saccule for the diagnosis of endolymphatic hydrops in Meniere disease, using a three-dimensional T2-weighted steady state free precession sequence: accurate, fast, and without contrast material intravenous injection. Eur Radiol Exp. 2017;1(1):14. doi: 10.1186/s41747-017-0020-7. Epub 2017 Oct 9. PMID 29708183
- [Background] Simon F, Guichard JP, Kania R, Franc J, Herman P, Hautefort C. Saccular measurements in routine MRI can predict hydrops in Meniere's disease. Eur Arch Otorhinolaryngol. 2017 Dec;274(12):4113-4120. doi: 10.1007/s00405-017-4756-8. Epub 2017 Sep 26. PMID 28951962
- [Derived] Connor S, Lally P, Pai I, Brnawi H, Touska P, Ourselin S, Hajnal JV. 7-Tesla sodium magnetic resonance imaging of the inner ears in unilateral Meniere's disease and endolymphatic hydrops: an exploratory study. BMC Med Imaging. 2025 Nov 11;25(1):454. doi: 10.1186/s12880-025-01986-6. PMID 41219717